CLINICAL TRIAL: NCT03193424
Title: A Prospective, Open-label, Randomized Controlled Clinical Study of Apatinib Combined With Docetaxel in the Treatment of Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Apatinib Combined With Docetaxel in the Treatment of Advanced Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, FanQingxia, Director, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHEAD-HNP001
Record Dates: First submitted 2017-06-17; First posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Advanced Esophageal Squamous Carcinoma
MeSH Terms: interventions — apatinib; Docetaxel

STUDY DESIGN:
Intervention Model Description: Double Group Assignment,apatinib plus docetaxel comparison to docetaxel.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib (Experimental)
  Interventions: Drug: Apatinib
- docetaxel (Active Comparator)
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Subjects were randomly divided into two groups,A group:apatinib 500mg/d,po,qd, Docetaxel 75 mg / m2 was administered on day 1 repeated every 21 days until progressive Disease(PD) . B group:Docetaxel 75 mg / m2 was administered on day 1 repeated every 21 days until progressive Disease(PD) .
  Other Names: Docetaxel

SUMMARY:
Esophageal cancer is a common malignant tumor in china, occupies the second place of malignant tumor morbidity and mortality, the overall 5-year survival rate less than 20%.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years old to 75 years old, male and female is ok.
* Esophageal squamous cell carcinoma diagnosed by histopathology and immunohistochemistry. At least one treated measurable lesion (spiral CT scan length ≥10mm, in line with RESCIST version 1.1 standard requirements);
* Patients with advanced esophageal cancer treated by radiotherapy and treatment;
* ECOG PS Rating: 0-1 points;
* Expected survival ≥12 weeks;
* Without molecular targeted drug therapy.
* The main organ function is normal, that is to meet the following criteria:

Blood test:a.HB≥90 g/L；b.ANC≥1.5×109/L；c.PLT ≥80×109/L； Biochemical tests:a.ALB≥30g / L；b. ALT和AST<2ULN；ALT and AST <2ULN;c.TBIL≤1.5ULN；Plasma Cr ≤ 1.5ULN;

* Subjects volunteered to join the study, signed informed consent, compliance, with follow-up.
* Researchers believe that patients can benefit.

Exclusion Criteria:

* Patients who have been confirmed to be allergic to apatinib and / or its excipients;
* Patients with uncontrollable hypertension (systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg, despite optimal drug therapy), with grade Ⅱ myocardial ischemia or myocardial infarction, poor control of arrhythmias (including QTc interval male ≥ 450 ms, female ≥470 ms).According to NYHA standard, grade Ⅲ ~ Ⅳ heart failure, or cardiac color Doppler ultrasound examination showed left ventricular ejection fraction (LVEF) <50%.
* Patients with a clear tendency to gastrointestinal bleeding, including the following: localized ulcer lesions, and fecal occult blood (++) can not be grouped; 2 months with black, hematemesis history;
* Coagulation dysfunction (INR> 1.5, APTT> 1.5 ULN), with bleeding tendency;
* (Eg, no swallowing, nausea, vomiting, chronic diarrhea and intestinal obstruction, etc.) that affect the absorption of oral medications;
* The patients with active brain metastases(without medical control) , cancer meningitis, spinal cord compression, or screening of imaging CT or MRI examination found that the brain or pia mater disease (21 days before the completion of treatment and symptoms of stable brain Metastasis patients can be grouped, but the need for transcranial MRI, CT or intravenous angiography, confirmed as no cerebral hemorrhage symptoms)
* Pregnant or lactating women
* Subject with other malignancies within 5 years(except the skin basal cell carcinoma and cervical in situ cancer that have already cured )
* Subject with a history of psychiatric abuse and who can not be abused or have mental disorders;
* Subject who participated in other drug clinical trials within 4 weeks.
* Subject who have received VEGFR inhibitors such as sorafenib, sunitinib;
* According to the investigator's judgment, there are serious illnesses that compromise the patient's safety or affect the patient's completion of the study;
* Researchers think it is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 6 months
  The first day of treatment to the date that disease progression is reported.

SECONDARY OUTCOMES:
Total Survival (OS) | up to 24 months
  the first day of treatment to death or last survival confirm date

CONTACTS AND LOCATIONS:
Locations (1):
- FirstAHZhengzhouU, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No